CLINICAL TRIAL: NCT02140658
Title: Affect of Multiple Health Education Interventions on Statins Medication Persistence and ClinicaL Prognosis of Ischemic Stroke Patients (HELP): a Prospective Cohort Study
Brief Title: Affect of Health Education on Statins Medication Persistence and ClinicaL Prognosis of Ischemic Stroke Patients (HELP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: yongjun wang (Other Government)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor-Investigator, yongjun wang, Professor,Vice president of Beijing Tiantan Hospital, Ministry of Science and Technology of the People´s Republic of China
Organization: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TTYY20140312
Record Dates: First submitted 2014-05-05; First posted 2014-05-16 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; Statins Medication Persistence; outcome
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multiple health education interventions (Active Comparator): The first group will receive health education manuals and Digital Video Disc (DVD) during hospitalization and regular health education messages during 6 months after discharge.
  Interventions: Behavioral: multiple health education interventions
- conventional health education (Placebo Comparator): The second group will receive conventional health education during hospitalization except health education manuals, regular health education messages and Digital Video Disc (DVD)
  Interventions: Behavioral: conventional health education

INTERVENTIONS:
Behavioral: multiple health education interventions
  Arms: multiple health education interventions
Behavioral: conventional health education
  Arms: conventional health education

SUMMARY:
The purpose of this study is to assess the affect of multiple health education interventions for statins medication Persistence and clinical prognosis of ischemic stroke patients at 3, 6 and 12 months.

DETAILED DESCRIPTION:
The study is a prospective, multicenter, hospital-based study on secondary prevention for patients with ischemic cerebrovascular diseases between May 2014 and June 2015. Physicians from 24 hospitals in Beijing underwent a standard secondary prevention training of ischemic cerebrovascular diseases by professional training, instruction manuals, stratification management software. In order to improve the persistence of taking preventive secondary medicine, IS patients from these 24 hospitals received healthy education through manuals and Digital Video Disc about health education during hospitalization and acquired secondary preventive knowledge of ischemic cerebrovascular diseases through regular health education messages during 6 months after discharge. Patients with IS from other 6 hospitals were used as a control, and no such intervention was given to them.

Telephone follow-up was performed at 3 months, 6 months, and 1 year after the onset of cerebral infarction, during which the use of antiplatelet and statins drugs and recurrence of IS were recorded. Patients who took antiplatelet drugs or statins at three follow-ups were regarded as persistent antiplatelet drugs or statins taking within one year after the onset of the disease. The main prognostic indicator was the recurrence of IS and persistence of statins medication within 1 year, and the main purpose was to explore the impact of persistent statins use on IS recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (male or female ≥18 years);
2. Acute ischemic stroke occured within 14 days of symptoms onset
3. Blood low density lipoprotein (LDL) ≧100mg/dl（2.59mmol/L）
4. Patients were prescribed statins at discharge
5. Patients signed informed consent
6. Patients have a cell phone and have the ability to receive and view messages

Exclusion Criteria:

1. Non-cerebrovascular events or hemorrhagic stroke
2. Patients have serious heart, liver, kidney dysfunction or coagulation disorders
3. Patients have circumstances that may affect the follow-up such as disturbance of consciousness, severe depression or other mental disorders, aphasia
4. Modified Rankin Scale score at discharge ≥3
5. Patients with severe vision or vision field impairment which may affect patients to read message in cell phone
6. Those who are participating in other clinical trials
7. Those who can not guarantee with the completion of 6 month follow-up after enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3111 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who continued taking statins drugs at three months after stroke onset. | 3 months after stroke onset
  Statins Medication persistence at 3 months. Patients who took statins at three months follow-up were regarded as persistent during three months.
Proportion of patients who continued taking statins drugs at six months after stroke onset. | 6 months after stroke onset
  Statins Medication persistence at 6 months.Patients who took statins at six months follow-up were regarded as persistent at six months.
Proportion of patients who continued taking statins drugs at 12 months after stroke onset. | 12 months after stroke onset
  Statins Medication persistence at 12 months.Patients who took statins at twelve months follow-up were regarded as persistent at twelve months.
Proportion of patients who continued taking statins drugs in 1 year after stroke onset. | 1 year after stroke onset
  Statins Medication persistence in 1 year: Patients who took statins at 3, 6 and 12 months follow-up were regarded as persistent during one year after stroke onset.
Recurrence of ischemic stroke in three months after stroke onset | 3 months after stroke onset
  Recurrence of ischemic stroke was defined as a new focal neurological deficit of vascular origin lasting >24 hours and without hemorrhage on computed tomography or MRI of the brain.
Recurrence of ischemic stroke in six months after stroke onset | 6 months after stroke onset
  Recurrence of ischemic stroke was defined as a new focal neurological deficit of vascular origin lasting >24 hours and without hemorrhage on computed tomography or MRI of the brain.
Recurrence of ischemic stroke in 12 months after stroke onset | 12 months after stroke onset
  Recurrence of ischemic stroke was defined as a new focal neurological deficit of vascular origin lasting >24 hours and without hemorrhage on computed tomography or MRI of the brain.

SECONDARY OUTCOMES:
Percentage of patients with 3-month poor clinical prognosis (including Death or Nonfatal myocardial infarction or Nonfatal hemorrhagic stroke or Severe disabilities) as a cluster and evaluated individually | 3 months after stroke onset
  Death included Vascular death and non-vascular death; Severe disabilities was defined as modified Rankin Scale ≥4
Percentage of patients with 6-month poor clinical prognosis (including Death or Nonfatal myocardial infarction or Nonfatal hemorrhagic stroke or Severe disabilities) as a cluster and evaluated individually | 6 months after stroke onset
  Death included Vascular death and non-vascular death; Severe disabilities was defined as modified Rankin Scale ≥4
Percentage of patients with 12-month poor clinical prognosis (including Death or Nonfatal myocardial infarction or Nonfatal hemorrhagic stroke or Severe disabilities) as a cluster and evaluated individually | 12 months after stroke onset
  Death included Vascular death and non-vascular death; Severe disabilities was defined as modified Rankin Scale ≥4

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082